CLINICAL TRIAL: NCT04636554
Title: Expanded Access Study of Phage Treatment in Covid-19 Patients on Anti-Microbials for Pneumonia or Bacteremia/Septicemia Due to A. Baumannii, P. Aeruginosa or S. Aureus
Brief Title: Personalized Phage Treatment in Covid-19 Patients With Bacterial Co-Infections Microbials for Pneumonia or Bacteremia/Septicemia
Status: No longer available | Type: Expanded Access
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: APT.APS.001
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Bacteremia; Septicemia; Acinetobacter Baumannii Infection; Pseudomonas Aeruginosa Infection; Staph Aureus Infection
Keywords: Covid19; Bacteriophage; Phage; Bacteremia; Septicemia; Acinetobacter; baumannii; Pseudomonas; Aeruginosa; Infection; Staph; Aureus
MeSH Terms: conditions — COVID-19; Bacteremia; Sepsis; Pseudomonas Infections; Infections; Staphylococcal Infections | interventions — Phage Therapy

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Other: Phage Therapy — Personalized intravenous phage therapy in Covid-19 patients along with anti-microbial treatment for pneumonia, bacteremia or septicemia due to A. baumannii, P. aeruginosa or S. aureus.

SUMMARY:
Phage Treatment in Covid-19 Patients with Bacterial Co-Infections

DETAILED DESCRIPTION:
The treatment approach will be to make phage therapy available to institutions who care for Covid-19 patients with bacterial co-infections due to A. baumannii, P. aeruginosa or S. aureus. Patient bacterial isolates will be tested to determine phage susceptibility prior to and during phage therapy.

The primary objectives are to determine the feasibility of developing, producing and providing a personalized intravenous phage for Covid-19 patients who have pneumonia, bacteremia or septicemia due to A. baumannii, P. aeruginosa or S. aureus and to evaluate the safety of intravenous phage in Covid-19 patients along with anti-microbial treatment for pneumonia, bacteremia or septicemia due to A. baumannii, P. aeruginosa or S. aureus.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 patients with pneumonia or bacteremia/septicemia who have culture-confirmed bacterial co-infection with A. baumannii, P. aeruginosa or S. aureus.
* Patient provided informed and signed consent.

Exclusion Criteria:

* Patient eligible for another APT sponsored trial.
* Patient participating in another clinical trial at the same time or patients < 4 weeks from participating in an alternative investigational protocol/study
* Patient with known allergy to infusion of phage products
* Patients with a history of Meningitis or encephalitis at time of study entry, Primary immune deficiency disease or tuberculosis or Stroke, transient ischemic attack (TIA), or untreated deep vein thrombosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult